CLINICAL TRIAL: NCT01204307
Title: A Phase III Study to Investigate the Differential Influence of Prior Chemotherapy on the Efficacy of Erlotinib in Patients With Advanced Non-small Cell Lung Cancer (IIIB, IV) With or Without EGFR Gene Mutation
Brief Title: Influence of Prior Chemotherapy on Clinical Benefit With Erlotinib in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer With or Without EGFR Gene Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Taiwan Chest Disease Association (Other)
Responsible Party: Principal Investigator, Chung Fu-Tsai, Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-1896C
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2010-09

CONDITIONS: Advanced Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Docetaxel; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- docetaxel/cisplatin (Experimental): The treatment schedule comprises a maximum of six 3-week treatment cycles consisting of weekly docetaxel (30 mg/m2) and cisplatin (37.5 mg/m2) for 2 consecutive weeks followed by a 1-week treatment-free period. The patients will be assessed after each cycle and a final assessment will be done after three and six cycles.
  Interventions: Drug: Docetaxel/cisplatin
- Pemetrexed/cisplatin (Active Comparator): The patients are given pemetrexed (500 mg/m2 as a 10-min intravenous infusion) and cisplatin (75 mg/m2) on day 1 every 21 days. Dexamethasone (4 mg) is administered twice daily on the day before, the day of, and the day after each dose of pemetrexed. Oral folic acid supplementation (1000 mg) is administered daily, beginning approximately 2 weeks prior to the first dose of pemetrexed and continues until 3 weeks after treatment discontinuation. A 1000 mg vitamin B12 injection is administered intramuscularly approximately 1-2 weeks before the first dose of pemetrexed and is repeated approximately every 9 weeks until 3 weeks after therapy discontinuation.
  Interventions: Drug: Pemetrexed/cisplatin

INTERVENTIONS:
Drug: Docetaxel/cisplatin — The treatment schedule comprises a maximum of six 3-week treatment cycles consisting of weekly docetaxel (30 mg/m2) and cisplatin (37.5 mg/m2) for 2 consecutive weeks followed by a 1-week treatment-free period. The patients will be assessed after each cycle and a final assessment will be done after three and six cycles.
  Other Names: Taxotere- made by Sanofi-Aventis.
  Arms: docetaxel/cisplatin
Drug: Pemetrexed/cisplatin — The patients are given pemetrexed (500 mg/m2 as a 10-min intravenous infusion) and cisplatin (75 mg/m2) on day 1 every 21 days. Dexamethasone (4 mg) is administered twice daily on the day before, the day of, and the day after each dose of pemetrexed. Oral folic acid supplementation (1000 mg) is administered daily, beginning approximately 2 weeks prior to the first dose of pemetrexed and continues until 3 weeks after treatment discontinuation. A 1000 mg vitamin B12 injection is administered intramuscularly approximately 1-2 weeks before the first dose of pemetrexed and is repeated approximately every 9 weeks until 3 weeks after therapy discontinuation.
  Other Names: Alimta- made by LiLy.
  Arms: Pemetrexed/cisplatin

SUMMARY:
To compare the differential influence of 1st line doublet chemotherapy containing Docetaxel versus Pemetrexed on clinical efficacy of Erlotinib as a second line therapy in patients with relapsed or progressed non-squamous NSCLC.

DETAILED DESCRIPTION:
The clinical management of advanced non-small cell lung cancer (NSCLC) remains challenging. Initial therapies for advanced NSCLC with platinum-based regimens have shown consistent overall response rates of 30% to 40% with progression-free intervals of 4-5 months and 1-year survival rates of 35% to 40% [1-3]. First line doublet chemotherapy commonly used in daily practice includes Gemcitabine, vinorelbine, paclitaxel and docetaxel those have proven efficacy with platinum against best supportive care, prolonging survival for approximately 3 months. Recently, pemetrexed, a multi-target antifolate agent, has been introduced into the 1st line doublet chemotherapy with platinum-based regimen to have similar efficacy and a better safety profile compared to docetaxel or gemcitabine [4]. Although those agents seem to have equivalent efficacy, tolerability tends to be a concern for docetoxel.

Myelosuppression with the standard docetaxel schedule of 75 mg/m2 administered once every 3 weeks is extremely frequent and severe; neutropenia occurs in 54% to 67% of patients and febrile neutropenia occurs in 1.8% to 8.0% of patients [5, 6]. Moreover, non-hematologic toxicities, such as grade 3-4 asthenia (12% to 18%), and nausea and vomiting (1% to 3.6%), are not uncommon [5, 6]. To increase tolerability of docetaxel, alternative schedules have been extensively studied. Accumulating evidence suggests that a weekly schedule of docetaxel (35 mg/m2) reduces severe and febrile neutropenia without decreasing antitumor activity [7-10]. Nevertheless, no significant differences were observed for anemia, thrombocytopenia, and non-hematologic toxicity [7]. For the same reason, a lower dose of docetaxel (60 mg/m2 every 3 weeks) has been recommended in Japan [11, 12]. However, recent large scale trials with such a dose of docetaxel still revealed high incidences of grade 3 and 4 neutropenia (up to 82.9%) [12-14]. Different schedules of low dose docetaxel have not been studied, nor has a comparison been made between low dose docetaxel and the less toxic agent, pemetrexed.

Currently, the investigators have been following a schedule of weekly low dose docetaxel (30 mg/m2 on days 1 and 8 every 3 weeks; 60 mg/m2 accumulated dose for each cycle) at our hospital in an effort to achieve better tolerability (in press-chemotherapy 2010). The investigators therefore perform an exploratory study, by prospective analysis, to investigate the efficacy and toxicity of such a low dose docetaxel schedule compared to that of pemetrexed in patients with NSCLC who are chemotherapy naive.

Erlotinib, an orally-available epidermal growth factor receptor (EGFR) tyrosine-kinase inhibitor (TKI), significantly prolongs survival and produces significant symptom and quality-of-life benefits compared with best supportive care in unselected patients with relapsed non-small-cell lung cancer (NSCLC) [15, 16]. In a large, phase III, placebo-controlled study (BR.21), erlotinib produced a survival benefit across all patient sub-groups studied [15].

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years, <75 years old
2. Pathological confirmation of non-squamous NSCLC
3. Clinical stage IIIB or IV
4. Measurable tumor size by RECIST criteria
5. ECOG <2
6. Adequate hematological laboratory parameters
7. Adequate hepatic, renal laboratory parameters

Exclusion Criteria:

1. Un-specified NSCLC
2. Prior therapy with any chemotherapy or EGFR TKI or monoclonal antibodies
3. Any unstable systemic disease (active infection, hypertension, unstable angina, CHF, liver cirrhosis, end stage renal failure etc., )
4. Nursing or pregnant mothers
5. Untreated Brain metastasis
6. ECOG>2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Response rate to erlotinib with Docetaxel/cisplatin or Pemetrexed/cisplatin | 2-3 months
  Eligible patients will be randomized to receive 1st line chemotherapy with either Docetaxel (60mg/m2)/Cisplatin (75mg/m2) or Pemetrexed (500mg/m2)/Cisplatin (75mg/m2) for 4-6 cycles. Patients will be followed up without any maintenance treatment after 4-6 cycles of chemotherapy.
  Once patients are found tumor relapse or in progression, all the patients will be prescribed Erlotinib 150 mg/day until disease progression, unacceptable toxicity or death. Patients will be followed up every 2-3 months for their responsive rate.

SECONDARY OUTCOMES:
Progression-free survival and overall survival after erlotinib treatment with 1st line Docetaxel/cisplatin or Pemetrexed/cisplatin. | 12-24 months
  Erlotinib 150 mg daily will be given to patients who are in progression after 1st line cisplatin-base doublet chemotherapy. Treatment will continue until documented disease progression, or patient refusal to continue. The progression-free survival encompasses the time from the start date of the Erlotinib treatment to documented progression, or death from any cause. The Overall survival from each arm of treatment is calculated from the start date of the treatment to death or to the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Han-Pin Kuo, MD, PhD, Study Director — Taiwan Chest Disease Association and Chang Gung Memorial Hospital
Locations (4):
- Taiwan (4):
  - Chang Gung Memorial Hospital, Taipei, Taipei
  - Chang Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - McKay Memorial Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei

REFERENCES:
- [Derived] Feng PH, Lee KY, Chang YL, Chan YF, Kuo LW, Lin TY, Chung FT, Kuo CS, Yu CT, Lin SM, Wang CH, Chou CL, Huang CD, Kuo HP. CD14(+)S100A9(+) monocytic myeloid-derived suppressor cells and their clinical relevance in non-small cell lung cancer. Am J Respir Crit Care Med. 2012 Nov 15;186(10):1025-36. doi: 10.1164/rccm.201204-0636OC. Epub 2012 Sep 6. PMID 22955317